CLINICAL TRIAL: NCT05067907
Title: Efficacy of Respiratory Physiotherapy on Severe ICU-admitted COVID-19 Patients: a Multicentric, National, Observational, Retrospective Study.
Brief Title: Efficacy of Respiratory Physiotherapy on Severe ICU-admitted COVID-19 Patients.
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: FISIO-UTI-COVID
Record Dates: First submitted 2021-08-30; First posted 2021-10-05 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: COVID-19 ICU-admitted patients that did not received physiotherapy interventions during ICU stay.
- Physiotherapy: COVID-19 ICU-admitted patients that received physiotherapy interventions during ICU stay.
  Interventions: Procedure: Early physiotherapy

INTERVENTIONS:
Procedure: Early physiotherapy — Respiratory physiotherapy included:
  1. early and functional mobilization: passive and active mobilization, muscle strengthening, improving independence in activities of daily living (ADL), sitting out of bed, standing, walking;
  2. patient positioning to achieve better ventilation/perfusion ratio and gas exchange;
  3. airway clearance;
  4. aerosol administration;
  5. invasive mechanical ventilation weaning;
  6. use of non-invasive mechanical ventilation (NIMV) and continuous positive airway pressure (CPAP);
  7. tracheostomy management and weaning;
  8. swallowing assessment;
  9. management of oxygen delivery;
  10. lung expansion;
  11. patient assessment and functional scale administration.
  Other Names: respiratory physiotherapy; early rehabilitation
  Groups: Physiotherapy

SUMMARY:
COVID-19 is an infectious disease caused by SARS-CoV2 virus. COVID-19 patients can develop a severe disease that can lead to hypoxic respiratory failure and acute respiratory distress syndrome (ARDS). Severe patients can require access to intensive care unit (ICU). Early rehabilitation is known to be effective in critically ill patients and in ARDS.

Early rehabilitation is known to be effective in critically ill subjects. The role of physiotherapy in severe COVID-19 patients is still unclear and few guidelines have been proposed so far. Aim of this study is to assess efficacy of early rehabilitation for severe ICU-admitted COVID-19 patients as compared to a group that did not received physiotherapy treatment in ICU.

DETAILED DESCRIPTION:
COVID-19 is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which emerged in China in December 2019 and in Italy in February 2020. A large proportion of infected people have mild clinical manifestations, whereas >10% develop a severe disease, which could evolve into acute hypoxemic respiratory failure (AHRF) and acute respiratory distress syndrome (ARDS) requiring intensive care unit (ICU) admission. A high proportion of ICU patients need invasive mechanical ventilation (IMV) and about 50% of the ICU-admitted patients die. The median age of ICU COVID-19 patients was <65 years and the mortality in patients aged <63 years ranges from 15 to 20%.

Early rehabilitation is safe and effective in critically ill patients and, in patients with ARDS, it helps to reduce the functional impairment due to the prolonged stay in ICU. Preliminary data suggest the implementation of early and active mobilization programs, as well as airway clearance, for patients with severe forms of COVID-19. To date, the role of respiratory physiotherapy in severe COVID-19 patients is still unclear.

Aim of this study is to assess efficacy of early rehabilitation for severe ICU-admitted COVID-19 patients as compared to a group that did not recevied physiotherapy treatment in ICU. Physiotherapy efficacy is evaluated in terms of ventilator free days (VFD) during the first 30 days after neuromuscular blockade stop.

Moreover, duration of ICU stay and patient functional status at ICU discharge will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having laboratory confirmed COVID-19 pneumonia
* Developed hypoxemic acute respiratory failure (hARF) requiring access to ICU
* Treated by physiotherapists during the ICU stay
* Stopped the neuromuscular blokade treatment

Exclusion Criteria:

* Previuos cognitive deficit (Mini menatal state examination <20)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will study patients accessing acute hospital ICU with hypoxemic acute respiratory failure (hARF) due to laboratory confirmed COVID-19 pneumonia form March 1st to May 30th.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days (VFD) and alive at day 28 | Up to 28 days after neuromuscular blokade stop
  To determine if early physiotherapy, as compared to no physiotherapy treatment, increases the number of ventilator-free days (VFD) and alive at day 28 in severe COVID-19 ICU-admitted patients.

SECONDARY OUTCOMES:
ICU stay duration | From ICU admission to ICU discharge; up to 60 days.
  Mean days of ICU stay
PaO2/FiO2 | At ICU discharge; up to 60 days
  Mean measure of PaO2/FiO2
ICU survival rate | From ICU admission until date of death from any cause, during ICU stay; up to 100 days.
  Number of patients that survived ICU stay
hospital survival rate | From ICU admission until date of death from any cause, during hospitalization
  Number of patients that survived hospitalization
90 days survival rate | From ICU admission until date of death from any cause, assessed up to 90 days after neuromuscular blokade removal
  Number of patients that survived during 90 days after neuromuscular blokade stop

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Privitera, MSC, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (4):
- Italy (4):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milan
  - Ospedale San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - APSS Provincia Autonoma di Trento Ospedale Santa Chiara, Trento

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Result] Kim RY, Murphy TE, Doyle M, Pulaski C, Singh M, Tsang S, Wicker D, Pisani MA, Connors GR, Ferrante LE. Factors Associated With Discharge Home Among Medical ICU Patients in an Early Mobilization Program. Crit Care Explor. 2019 Nov 11;1(11):e0060. doi: 10.1097/CCE.0000000000000060. eCollection 2019 Nov. PMID 32166241
- [Result] Lazzeri M, Lanza A, Bellini R, Bellofiore A, Cecchetto S, Colombo A, D'Abrosca F, Del Monaco C, Gaudiello G, Paneroni M, Privitera E, Retucci M, Rossi V, Santambrogio M, Sommariva M, Frigerio P. Respiratory physiotherapy in patients with COVID-19 infection in acute setting: a Position Paper of the Italian Association of Respiratory Physiotherapists (ARIR). Monaldi Arch Chest Dis. 2020 Mar 26;90(1). doi: 10.4081/monaldi.2020.1285. PMID 32236089
- [Derived] Privitera E, Gambazza S, Rossi V, Santambrogio M, Binda F, Tarello D, Caiffa S, Turrin V, Casagrande C, Battaglini D, Panigada M, Fumagalli R, Pelosi P, Grasselli G. Association of ventilator-free days with respiratory physiotherapy in critically ill patients with Coronavirus Disease 2019 (COVID-19) during the first pandemic wave. A propensity score-weighted analysis. Front Med (Lausanne). 2022 Sep 12;9:994900. doi: 10.3389/fmed.2022.994900. eCollection 2022. PMID 36172535